CLINICAL TRIAL: NCT06678425
Title: Efficacy of Repetitive Peripheral Magnetic Stimulation on Shoulder Subluxation in Subacute Stroke Patients
Brief Title: This Study is About the Efficacy of Repetitive Peripheral Magnetic Stimulation on the Treatment of Shoulder Subluxation in Subacute Stroke Patients.
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2024/673; Ramathibodi Hospital (Other: Ramathibodi Hospital)
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Shoulder Subluxation; Subacute Stroke; Magnetic Stimulation; Randomised Controlled Trial

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, Double-blind, Sham-controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real rPMS (Experimental): Real rPMS was applied to supraspinatus and posterior deltoid muscles for 20 Hz total 2,400 pulses.
  Interventions: Device: Peripheral magnetic stimulator
- sham rPMS (Sham Comparator): sham rPMS was applied to supraspinatus and posterior deltoid muscles with the same coil as real rPMS, but in a position perpendicular to the skin, using intensity for 5% of the maximum output.
  Interventions: Device: Peripheral magnetic stimulator

INTERVENTIONS:
Device: Peripheral magnetic stimulator — a non-invasive method of delivering a rapidly pulsed, high-intensity magnetic field to peripheral muscles
  Other Names: PMS
  Arms: real rPMS
Device: Peripheral magnetic stimulator — The same coil as real rPMS, but in a position perpendicular to the skin
  Other Names: PMS
  Arms: sham rPMS

SUMMARY:
The goal of this clinical trial is to study the efficacy of repetitive peripheral magnetic stimulation (rPMS) on shoulder subluxation in subacute stroke patients. The main questions it aims to answer are Could rPMS reduce shoulder subluxation and improve upper-limb motor recovery in subacute stroke patients?

Researchers will compare real rPMS to sham rPMS to see if rPMS works to improve shoulder subluxation and upper-limb motor recovery in subacute stroke patients.

Participants will:

* Get real rPMS or sham rPMS for 20 minutes, 5 days a week for 2 weeks
* Get conventional rehabilitation program 5 days a week for 2 weeks
* Follow-up at 2-, 4-, 8- and 12-weeks after first day of treatment

ELIGIBILITY:
Inclusion Criteria:

* Subacute phase (seven days to six months) and first time of stroke patients
* Shoulder subluxation that measured half of a fingerbreadth or more
* Meet the criteria for admission to a comprehensive rehabilitation program
* Medically stable
* Intact skin on the hemiparetic arm

Exclusion Criteria:

* Patients with contraindication for magnetic stimulation; cardiac pacemakers, magnetic materials near the intended stimulation site
* Patients with pregnancy
* Patients with severe aphasia or severe cognitive impairment
* Patients with previous shoulder pathology or limit shoulder function before stroke
* Patients with unstable vital signs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acromiohumeral interval | pretreatment, 2-, 4-, 8- and 12-weeks after first day of treatment
  the shortest distance between two parallel lines drawn from the inferior border of the acromion and the superior border of the humerus head on the anteroposterior shoulder x-ray

SECONDARY OUTCOMES:
Fugl-Meyer assessment of upper extremities (FMA-UE) | pretreatment, 2-, 4-, 8- and 12-weeks after first day of treatment
  a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. Maximum score for upper extremity is 66 points.
Modified Ashworth Scale (MAS) | pretreatment, 2-, 4-, 8- and 12-weeks after first day of treatment
  a grade of spasticity from a 0-4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch.
Numeric Pain Rating Scale (NRS) | pretreatment, 2-, 4-, 8- and 12-weeks after first day of treatment
  Measuring of pain intensity, respondents are asked to choose the single number that best represents their pain intensity, on a 0 (No Pain) to 10 (Worst pain) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hemrungrojn S, Tangwongchai S, Charoenboon T, Panasawat M, Supasitthumrong T, Chaipresertsud P, Maleevach P, Likitjaroen Y, Phanthumchinda K, Maes M. Use of the Montreal Cognitive Assessment Thai Version to Discriminate Amnestic Mild Cognitive Impairment from Alzheimer's Disease and Healthy Controls: Machine Learning Results. Dement Geriatr Cogn Disord. 2021;50(2):183-194. doi: 10.1159/000517822. Epub 2021 Jul 29. PMID 34325427
- [Result] Manigandan JB, Ganesh GS, Pattnaik M, Mohanty P. Effect of electrical stimulation to long head of biceps in reducing gleno humeral subluxation after stroke. NeuroRehabilitation. 2014;34(2):245-52. doi: 10.3233/NRE-131041. PMID 24419017
- [Result] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Result] Gladstone DJ, Danells CJ, Black SE. The fugl-meyer assessment of motor recovery after stroke: a critical review of its measurement properties. Neurorehabil Neural Repair. 2002 Sep;16(3):232-40. doi: 10.1177/154596802401105171. PMID 12234086
- [Result] Jiang YF, Zhang D, Zhang J, Hai H, Zhao YY, Ma YW. A Randomized Controlled Trial of Repetitive Peripheral Magnetic Stimulation applied in Early Subacute Stroke: Effects on Severe Upper-limb Impairment. Clin Rehabil. 2022 May;36(5):693-702. doi: 10.1177/02692155211072189. Epub 2022 Jan 5. PMID 34985366
- [Result] Hall J, Dudgeon B, Guthrie M. Validity of clinical measures of shoulder subluxation in adults with poststroke hemiplegia. Am J Occup Ther. 1995 Jun;49(6):526-33. doi: 10.5014/ajot.49.6.526. PMID 7645665
- [Result] Yang C, Chen P, Du W, Chen Q, Yang H, Su M. Musculoskeletal Ultrasonography Assessment of Functional Magnetic Stimulation on the Effect of Glenohumeral Subluxation in Acute Poststroke Hemiplegic Patients. Biomed Res Int. 2018 Jul 3;2018:6085961. doi: 10.1155/2018/6085961. eCollection 2018. PMID 30065941
- [Result] Fujimura K, Kagaya H, Endou C, Ishihara A, Nishigaya K, Muroguchi K, Tanikawa H, Yamada M, Kanada Y, Saitoh E. Effects of Repetitive Peripheral Magnetic Stimulation on Shoulder Subluxations Caused by Stroke: A Preliminary Study. Neuromodulation. 2020 Aug;23(6):847-851. doi: 10.1111/ner.13064. Epub 2019 Nov 5. PMID 32840021
- [Result] Beaulieu LD, Schneider C. Effects of repetitive peripheral magnetic stimulation on normal or impaired motor control. A review. Neurophysiol Clin. 2013 Oct;43(4):251-60. doi: 10.1016/j.neucli.2013.05.003. Epub 2013 Jun 10. PMID 24094911
- [Result] Linn SL, Granat MH, Lees KR. Prevention of shoulder subluxation after stroke with electrical stimulation. Stroke. 1999 May;30(5):963-8. doi: 10.1161/01.str.30.5.963. PMID 10229728
- [Result] Stecker MM, Patterson T, Netherton BL. Mechanisms of electrode induced injury. Part 1: theory. Am J Electroneurodiagnostic Technol. 2006 Dec;46(4):315-42. PMID 17285816
- [Result] Lee JH, Baker LL, Johnson RE, Tilson JK. Effectiveness of neuromuscular electrical stimulation for management of shoulder subluxation post-stroke: a systematic review with meta-analysis. Clin Rehabil. 2017 Nov;31(11):1431-1444. doi: 10.1177/0269215517700696. Epub 2017 Mar 27. PMID 28343442
- [Result] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Result] Arya KN, Pandian S, Puri V. Rehabilitation methods for reducing shoulder subluxation in post-stroke hemiparesis: a systematic review. Top Stroke Rehabil. 2018 Jan;25(1):68-81. doi: 10.1080/10749357.2017.1383712. Epub 2017 Oct 11. PMID 29017429
- [Result] Adey-Wakeling Z, Liu E, Crotty M, Leyden J, Kleinig T, Anderson CS, Newbury J. Hemiplegic Shoulder Pain Reduces Quality of Life After Acute Stroke: A Prospective Population-Based Study. Am J Phys Med Rehabil. 2016 Oct;95(10):758-63. doi: 10.1097/PHM.0000000000000496. PMID 27003204
- [Result] Kumar P, Fernando C, Mendoza D, Shah R. Risk and associated factors for hemiplegic shoulder pain in people with stroke: a systematic literature review. Physical Therapy Reviews. 2021;27(3):191-204.
- [Result] Paci M, Nannetti L, Taiti P, Baccini M, Rinaldi L. Shoulder subluxation after stroke: relationships with pain and motor recovery. Physiother Res Int. 2007 Jun;12(2):95-104. doi: 10.1002/pri.349. PMID 17536647
- [Result] Stolzenberg D, Siu G, Cruz E. Current and future interventions for glenohumeral subluxation in hemiplegia secondary to stroke. Top Stroke Rehabil. 2012 Sep-Oct;19(5):444-56. doi: 10.1310/tsr1905-444. PMID 22982832
- [Result] Suethanapornkul S, Kuptniratsaikul PS, Kuptniratsaikul V, Uthensut P, Dajpratha P, Wongwisethkarn J. Post stroke shoulder subluxation and shoulder pain: a cohort multicenter study. J Med Assoc Thai. 2008 Dec;91(12):1885-92. PMID 19133525
- [Result] Turner-Stokes L, Jackson D. Shoulder pain after stroke: a review of the evidence base to inform the development of an integrated care pathway. Clin Rehabil. 2002 May;16(3):276-98. doi: 10.1191/0269215502cr491oa. PMID 12017515
- [Result] Paci M, Nannetti L, Rinaldi LA. Glenohumeral subluxation in hemiplegia: An overview. J Rehabil Res Dev. 2005 Jul-Aug;42(4):557-68. doi: 10.1682/jrrd.2004.08.0112. PMID 16320150